CLINICAL TRIAL: NCT02091193
Title: Effects of Krill Oil on Endothelial Function in Patients With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Danbury Hospital (Other)
Collaborators: Prograde Nutrition (Unknown)
Responsible Party: Principal Investigator, Joann Petrini, PhD, MPH, Director, Clinical and Health Outcomes Research, Danbury Hospital
Other Study IDs: 12-02-34-334
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Type II Diabetes Mellitus
Keywords: Krill Oil; Endothelial Function; Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Only serum is retained and is discarded after specified assays are completed. No analysis requires genetic information.

GROUPS / COHORTS (2):
- Placebo to Krill Oil: Group 2 receives supplement B for four weeks, undergoes a two week washout period, and then receives supplement A for another four weeks. Measurements are taken at baseline, after supplement B completion and after supplement A completion. Participants are informed which supplement was krill oil and which was placebo following completion of this phase of the study. Group 2 participants are given an option to also take an additional 17 weeks of Krill Oil and return for a follow up evaluating the long term use of krill oil.
  Interventions: Dietary Supplement: Krill Oil (Supplement A); Dietary Supplement: Placebo (Supplement B)
- Krill Oil to Placebo: Group 1 receives supplement A for four weeks, undergoes a two week washout period, and then receives supplement B for another four weeks. Measurements are taken at baseline, after supplement A completion and after supplement B completion. Participants are informed which supplement was krill oil and which was placebo following completion of this phase of the study. Group 1 participants are given an option to also take an additional 17 weeks of Krill Oil and return for a follow up evaluating the long term use of krill oil.
  Interventions: Dietary Supplement: Krill Oil (Supplement A); Dietary Supplement: Placebo (Supplement B)

INTERVENTIONS:
Dietary Supplement: Krill Oil (Supplement A)
  Other Names: Prograde, Inc. Krill Oil
Dietary Supplement: Placebo (Supplement B)

SUMMARY:
The purpose of this study is to evaluate the effects of krill oil supplementation in patients with Type 2 diabetes mellitus on heart health and laboratory diabetic measurements.

Patients who enroll in this study will be asked to visit the Western Connecticut Health Network Biomedical Research Institute on 3 separate occasions: for baseline testing, after 4 weeks of supplementing with krill oil, and after 4 weeks of supplementing with a placebo. Patients will be randomized into one of two groups to determine the order in which they receive the supplement and placebo. Every patient will receive both the krill oil and the placebo, but both the coordinator and the patient are blinded to which is which. At each visit, participants will undergo a non-invasive test which measures the function of the inner lining of blood vessels and they will also have blood drawn. Fasting is required before each appointment. The blood drawn is used to measure their Hemoglobin A1C, Glucose, HDL, LDL, total cholesterol, C-peptide and total antioxidant capacity.

Risks to taking krill oil supplements are likely to include bad breath, heartburn, fishy taste, upset stomach, nausea, loose stools, gas, and bloating. Risks of EndoPAT testing are not permanent and may include pain, numbness, tingling, redness, and bruising at the site of the blood pressure cuff. Risks that are associated with drawing blood may include redness, swelling, pain or discomfort, bruising at the site of the needle stick, or in very rare cases, infection at the needle site. To minimize these risks, trained technologists and phlebotomists will be used for all procedures.

This is not a treatment option; while involved in this study all participants will continue their regular treatment for Type 2 diabetes mellitus (as well as any other applicable conditions).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 2 Diabetes Mellitus
* Stable on glucose lowering agents

Exclusion Criteria:

* Age of less than 18
* Currently pregnant or lactating
* Blood coagulation disorder or taking oral anticoagulants other than aspirin
* Seafood allergy
* Presently taking fish oil or krill oil supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The groups are selected from primary care offices, a diabetes and endocrine office, as well as self-referrals and medical record confirmed cases of Type 2 Diabetes Mellitus.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in Endothelial Function with Krill Oil Supplementation as Compared with Baseline and Placebo | Three Months

SECONDARY OUTCOMES:
Change in Lipid Profile (HDL, LDL, Total Cholesterol), Glucose, Hemoglobin A1C with Krill Oil Supplementation Compared with Baseline and Placebo | Three months

OTHER OUTCOMES:
Change C-Peptide and Total Antioxidant Capacity of Serum Compared with Baseline and Placebo | Three Months
Effects of Longer Term Krill Oil Supplementation compared to Baseline on Endothelial function, lipid profile, Hemoglobin A1C, glucose, c-peptide and total antioxidant capacity. | 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Ahmadi, MD, MPH, Principal Investigator — Danbury Hospital
Locations (1):
- Danbury Hospital, Danbury, Connecticut, United States

REFERENCES:
- [Background] Wijendran V, Huang MC, Diau GY, Boehm G, Nathanielsz PW, Brenna JT. Efficacy of dietary arachidonic acid provided as triglyceride or phospholipid as substrates for brain arachidonic acid accretion in baboon neonates. Pediatr Res. 2002 Mar;51(3):265-72. doi: 10.1203/00006450-200203000-00002. PMID 11861929
- [Background] Maki KC, Reeves MS, Farmer M, Griinari M, Berge K, Vik H, Hubacher R, Rains TM. Krill oil supplementation increases plasma concentrations of eicosapentaenoic and docosahexaenoic acids in overweight and obese men and women. Nutr Res. 2009 Sep;29(9):609-15. doi: 10.1016/j.nutres.2009.09.004. PMID 19854375
- [Background] Bunea R, El Farrah K, Deutsch L. Evaluation of the effects of Neptune Krill Oil on the clinical course of hyperlipidemia. Altern Med Rev. 2004 Dec;9(4):420-8. PMID 15656713
- [Background] Wong CY, Yiu KH, Li SW, Lee S, Tam S, Lau CP, Tse HF. Fish-oil supplement has neutral effects on vascular and metabolic function but improves renal function in patients with Type 2 diabetes mellitus. Diabet Med. 2010 Jan;27(1):54-60. doi: 10.1111/j.1464-5491.2009.02869.x. PMID 20121889
- [Derived] Lobraico JM, DiLello LC, Butler AD, Cordisco ME, Petrini JR, Ahmadi R. Effects of krill oil on endothelial function and other cardiovascular risk factors in participants with type 2 diabetes, a randomized controlled trial. BMJ Open Diabetes Res Care. 2015 Oct 14;3(1):e000107. doi: 10.1136/bmjdrc-2015-000107. eCollection 2015. PMID 26504524
- See also: Prograde, Inc Krill Oil Information — http://getprograde.com/essential-fatty-acid.html